CLINICAL TRIAL: NCT02348450
Title: Irinotecan Plus Cisplatin Compared With Etoposide Plus Cisplatin for Extensive Stage Small-cell Lung Cancer: a Multi-center, Randomized, Open Label Study
Brief Title: Irinotecan Plus Cisplatin Compared With Etoposide Plus Cisplatin for Extensive Stage Small-cell Lung Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1404
Record Dates: First submitted 2014-10-23; First posted 2015-01-28 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irinotecan plus Cisplatin (Experimental): first line: irinotecan 65mg/m2 d1,8. Cisplatin 30mg/m2，d1,8, 21days/cycle×6 cycles Second-line: etoposide alone OR etoposide plus cisplatin, dosage will be same as first line or on investigator's discretion.
  Interventions: Drug: Irinotecan; Drug: Cisplatin
- Etoposide plus Cisplatin (Experimental): first line: etoposide 60mg/m2 d1-5 Cisplatin 75mg/m2，d1(recommended), or administer three times with same total daily dose , 21days/cycle×6 cycles Second-line: irinotecan alone or irinotecan plus cisplatin, dosage is same as first line or on investigator's discretion.
  Interventions: Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: Irinotecan — 40mg
  Other Names: Ai Li
  Arms: Irinotecan plus Cisplatin
Drug: Etoposide — 5ml：0.1g
  Other Names: H32025583
  Arms: Etoposide plus Cisplatin
Drug: Cisplatin — 6ml：30mg
  Other Names: Nuo Xin

SUMMARY:
This study is aimed to evaluate the progression-free survival(PFS) and also survival of IP and EP (head-to-head) as the first line therapy for extensive stage small-cell lung cancer and to explore the reasonable first-line therapy for Chinese population. An open-label, multi-center study will be conducted with dynamic randomization of approximately 1:1 ratio with an estimation of 308 eligible participants.

DETAILED DESCRIPTION:
evaluate the progression-free survival(PFS) and also survival of IP and EP (head-to-head) as the first line therapy for extensive stage small-cell lung cancer and to explore the reasonable first-line therapy for Chinese population.

An open-label, multi-center study will be conducted with dynamic randomization of approximately 1:1 ratio with an estimation of 308 eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed extensive stage small-cell lung cancer (remote metastasis and/or contralateral lymph-node involvement; not those with simple ipsilateral pleural effusion);
* No prior radiotherapy, chemotherapy or surgery;
* At least one measurable lesion, CT≥20mm, spiral CT≥10mm(diameter);
* ECOG PS 0-1;
* Age 18-70;
* Life expectancy > three months;
* In general normal function of heart, liver, kidney and bone marrow;
* WBC C>4.0×10(9)/L, NEUT>1.50×10(9)/L, PLT>100×10(9)/L, Hb>95g/L;
* Liver function: TBIL < 1.5 x UL normal range; ALT and AST < 1.5 x UL normal range;
* Kidney function: normal serum creatinine level;
* Signed an informed consent and will comply with the study protocol and follow-up plans.

Exclusion Criteria:

* Failed to meet the entry criteria of pathology and clinical stage;
* Have received prior chemotherapy or target treatment;
* Currently receiving other anticancer therapy;
* No measurable lesions or lesions cannot be assessed;
* Patients with acute or chronic medical or psychiatric condition, or laboratory abnormalities that may impact the judgment of the investigator and the result of the study, determined by investigator they may include:

Uncontrolled tumor metastasis in central nerve system; Uncontrolled hypertension, unstable angina, MI history, or congestive heart-failure, uncontrolled arrhythmia, ischemic vascular disease within the 12 months prior to study treatment; Myocardial ischemia by ECG or valvular heart disease; Grade 3 or above peripheral neuropathy; Active stage of infection by bacteria, fungi or virus; Pregnant or breast feeding woman; History of uncontrolled mental disease.

* Not able to discontinue NSAIDs treatment;
* Other active malignant tumors except non-melanoma skin cancer, in-situ cervical carcinoma and cured early prostatic carcinoma;
* Patients with allergies, known or may be allergic to drugs in research;
* Patients with poor compliance to treatment and follow-up;
* Patients with UGT1A1-6 and UGT1A1-28 gene mutation;
* With clinical symptoms of brain metastasis(patient with stable clinical performance and no need to treat can be included in the trial);
* Chest, abdominal or pericardial effusion that needs anti-cancer intervention;
* Accompanied with Grade ≥2 diarrhea;
* Participated in other clinical trials within one month before randomization;
* Investigator's judgment to exclude.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival of first line therapy | 24 months

SECONDARY OUTCOMES:
Overall survival | 36 months
Objective Response Rate | 24 months
Number of patients experience adverse events | 36 months
Progression free survival of second line therapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D, Principal Investigator — Shanghai Chest hospital of Shanghai Jiaotong University
Locations (20):
- China (20):
  - The First Affiliated Hospital of AnHui Medical University, Hefei, Anhui
  - FuJian Provincial Tumor Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Cancer Hospital Affiliated To GuangXi Medical University, Nanning, Guangxi
  - Fourth hospital of hebei medical university, Shijiazhuang, Hebei
  - The First Affiliated Hospital of HaErBin Medical University, Haerbin, Heilongjiang
  - HeNan Provincial Tumor Hospital, Zhengzhou, Henan
  - WuHan Tongji Hospital, Wuhan, Hubei
  - HuNan Provincial Tumor Hospital, Changsha, Hunan
  - JiangSu Provincial Tumor Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - LiaoNing Provincial Tumor Hospital, Shenyang, Liaoning
  - ShanDong Provincial Tumor Hospital, Jinan, Shandong
  - Linyi cancer hospital, Linyi, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - East Hospital Affiliated To Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Chest hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang
  - ZheJiang Provincial Tumor Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No